CLINICAL TRIAL: NCT03400956
Title: A Randomized, Parallel-group, Double-blind and Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of Vilaprisan in Subjects With Uterine Fibroids
Brief Title: Assess Safety and Efficacy of Vilaprisan in Subjects With Uterine Fibroids (ASTEROID 4)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a change in the development program, the study was closed prematurely.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15790; 2016-003561-26 (EudraCT Number)
Record Dates: First submitted 2018-01-05; First posted 2018-01-17 (Actual); Results first posted 2021-04-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Uterine Fibroids
Keywords: Heavy menstrual bleeding
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — vilaprisan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vilaprisan (A1) (Experimental): Vilaprisan in treatment period 1 for 12 weeks and in treatment period 2 for 12 weeks, separated by 1 bleeding episode.
  Interventions: Drug: Vilaprisan (BAY1002670)
- Placebo+Vilaprisan (B1) (Experimental): Placebo in treatment period 1 for 12 weeks, and vilaprisan in treatment period 2 for 12 weeks, separated by 1 bleeding episode.
  Interventions: Drug: Vilaprisan (BAY1002670); Drug: Placebo
- Vilaprisan+Placebo (B2) (Experimental): Vilaprisan in treatment period 1 for 12 weeks, and placebo in treatment period 2 for 12 weeks, separated by 1 bleeding episode.
  Interventions: Drug: Vilaprisan (BAY1002670); Drug: Placebo

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — Orally, coated tablet 2 mg, once daily
Drug: Placebo — Orally, coated tablet, once daily
  Arms: Placebo+Vilaprisan (B1); Vilaprisan+Placebo (B2)

SUMMARY:
The primary objective of this study was to show superiority of vilaprisan in the treatment of heavy menstrual bleeding (HMB) in subjects with uterine fibroids compared to placebo

The secondary objectives of this study were to additionally evaluate the efficacy and safety of vilaprisan in subjects with uterine fibroids

ELIGIBILITY:
Inclusion Criteria:

* Women, 18 years or older in good general health
* Diagnosis of uterine fibroid(s) documented by ultrasound at screening with at least 1 fibroid with largest diameter more than 30 mm and less than 120 mm
* Heavy menstrual bleeding (HMB) in at least 2 bleeding periods during the screening period each with blood loss volume of >80.00 mL documented by the alkaline hematin (AH) method
* An endometrial biopsy performed during the screening period without significant histological disorder such as endometrial hyperplasia (including simple hyperplasia) or other significant endometrial pathology
* Use of an acceptable non-hormonal method of contraception (ie, either male condom, cap, diaphragm or sponge, each in combination with spermicide) starting at Visit 1 until the end of the study

Exclusion Criteria:

* Pregnancy or lactation (less than 3 months since delivery, abortion, or lactation before start of treatment)
* Hypersensitivity to any ingredient of the study drug
* Hemoglobin values ≤6 g/dL or any condition requiring immediate blood transfusion (subjects with hemoglobin values ≤10.9 g/dL will be recommended to use iron supplementation)
* Any diseases, conditions, or medications that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Abuse of alcohol, drugs or medicines (e.g. laxatives)
* Use of other treatments that might interfere with the conduct of the study or the interpretation of results
* Undiagnosed abnormal genital bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (87):
- United States (46):
  - Clearview Medical Research, LLC, Canyon Country, California
  - Diagnamics, Inc., Encinitas, California
  - National Research Institute, Huntington Park, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - West Coast OB/GYN Associates, La Mesa, California
  - National Research Institute, Panorama City, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Vital Pharma Research, Hialeah, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Genoma Research Group, Inc., Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Vista Health Research, Miami, Florida
  - Palmetto Professional Research, Miami, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - A Premier Medical Research of Florida, LLC, Orange City, Florida
  - Clinical Neurosciences Solutions, Inc. DBA CNS Healthcare, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - DMI Research, Pinellas Park, Florida
  - Physician Care Clinical Research, Sarasota, Florida
  - Journey Medical Research, Snellville, Georgia
  - Women's Healthcare Associates, PA, Idaho Falls, Idaho
  - New England Center for Clinical Research, Inc., Fall River, Massachusetts
  - Altea Research Institute, Las Vegas, Nevada
  - Unified Women's Clinical Research, Greensboro, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Unified Women's Clinical Research / Ocala, FL, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vista Clinical Research, Columbia, South Carolina
  - Chattanooga Women for Women, Hixson, Tennessee
  - Women Partners in Health Obstetrics & Gynecology (OB/GYN), Austin, Texas
  - Gadolin Research, Beaumont, Texas
  - Discovery Clinical Trials, Dallas, Texas
  - Advances in Health, Inc., Houston, Texas
  - Discovery Clinical Trials, San Antonio, Texas
  - Center of Reproductive Medicine, Webster, Texas
  - Tidewater Physicians for Women, Norfolk, Virginia
  - Seattle Clinical Research Center, Seattle, Washington
- Czechia (5):
  - GynPorCentrum s.r.o., Krnov
  - Gynekologie MUDr. Jaromir Karban s.r.o, Neratovice
  - Privatni gynekologicko-porodnicka ordinace, Prague
  - GYNEVI s.r.o., Rokycany
  - Gynekologicka ambulance - Zabreh na Morave, Zábřeh
- Japan (26):
  - Funabashi Municipal Medical Center, Funabashi, Chiba
  - Tsujinaka Hospital Kashiwanoha, Kashiwa, Chiba
  - Matsudo City General Hospital, Matsudo, Chiba
  - Hashimoto Clinic, Sapporo, Hokkaido
  - Ena Odori Clinic, Sapporo, Hokkaido
  - Tokeidai Memorial Clinic, Sapporo, Hokkaido
  - Yoshio Clinic, Sapporo, Hokkaido
  - Kosumo Clinic, Kako-gun, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Asahi-Clinic., Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa
  - Kyoto city Hospital, Nakagyo-ku, Kyoto
  - Medical Topia Soka Hospital, Sōka, Saitama
  - Omi Medical Center, Kusatsu, Shiga
  - Saiseikai Fukuoka General Hospital, Fukuoka
  - Unoki Clinic, Kagoshima
  - Tetsu-Nakamura Obstetrics and Gynecology Internal Medicine, Kagoshima
  - Four Seasons Ladies' Clinic, Kumamoto
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Ijinkai Takeda General Hospital, Kyoto
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - Gokeikai Osaka Kaisei Hospital, Osaka
  - Osaka City Hospital Organization Osaka City General Hospital, Osaka
  - Medical Co. LEADING GIRLS Women's Clinic LUNA Shinsaibashi, Osaka
- Russia (7):
  - Altai State Medical University, Barnaul
  - Maternity Hospital, 17, Saint Petersburg
  - Med Estetic Center, Saint Petersburg
  - "Granti-Med", Saint Petersburg
  - Scien. Res. Institute of Obsterics, Gyn. & Reproduction, Saint Petersburg
  - Close Joint Stock Company "Medical Company IDK", Samara
  - Smolensk State Medical University, Smolensk
- Ukraine (3):
  - Chernivtsi Regional Perinatal Center, Chernivtsi
  - Vinnytsia City Clinical Maternity Hospital No 2, Vinnytsia
  - Zaporizhzhia Regional Clinical Hospital, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — https://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 87 study centers in USA, Japan, Czech Republic, Russia, and Ukraine between 24-Jan-2018 (first participant first visit) and 30-Jun-2021 (last participant last visit).
Pre-assignment Details: Overall, 481 participants were screened, of them, 378 (78.6%) participants were not randomized to treatment. The majority of these (n=286) were screen failures. Of the 103 participants who were randomized, 91 participants received study treatment. Full analysis set (FAS) consisted of all randomized subjects, excluding randomized subjects who did not start treatment period 1 (never received study drug) due to the study being closed prematurely (7 [6.8%]), and included 96 (93.2%) subjects.
Groups:
- Vilaprisan (A1): Vilaprisan in treatment period (TP) 1 for 12 weeks and in treatment period 2 for 12 weeks, separated by 1 bleeding episode.
Period: Treatment Period 1
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Started (Allocated) | 35 | 34 | 34
Treated | 31 | 30 | 30
FAS (Full analysis set) | 32 | 33 | 31
Completed | 31 | 26 | 25
Not Completed | 4 | 8 | 9
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Study terminated by sponsor | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 4
Not completed — Other | 1 | 2 | 3
Period: Post-treatment Period 1
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Started | 31 | 26 | 25
Completed | 9 | 10 | 9
Not Completed | 22 | 16 | 16
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Physician Decision | 2 | 3 | 0
Not completed — Study terminated by sponsor | 11 | 10 | 11
Not completed — Withdrawal by Subject | 5 | 0 | 0
Not completed — Other | 4 | 3 | 4
Period: Treatment Period 2
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Started (Treatment started) | 9 | 10 | 9
Completed | 5 | 7 | 5
Not Completed | 4 | 3 | 4
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Other | 1 | 1 | 0
Period: Follow-up Period
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Started | 6 | 9 | 7
Completed | 6 | 9 | 5
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants in Full analysis set (FAS) was analyzed. The FAS consisted of all randomized subjects, excluding randomized subjects who did not start treatment Period 1 (never received study drug) due to the study being temporarily paused, including 96 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2) | Total
Number analyzed (Participants) | 32 | 33 | 31 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (5.5) | 42.7 (6.0) | 43.8 (4.3) | 43.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 31 | 96
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5 | 10
  Not Hispanic or Latino | 30 | 30 | 26 | 86
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 11 | 11 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 8 | 21
  White | 13 | 15 | 10 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 4
Endometrial thickness [Mean (Standard Deviation); unit: Millimeters] — Ultrasound examinations were performed. Endometrial thickness was measured in the medio-sagittal section as double-layer in millimeters. Baseline data of endometrial thickness is provided in below table. Population: Safety analysis set (SAF) was analyzed. The SAF consisted of all randomized participants who took at least 1 dose of study drug and included 91 (88.3%) participants.
  Millimeters
    number analyzed (Participants) | 31 | 30 | 30 | 91
    (all) | 12.8 (4.5) | 12.8 (2.9) | 11.9 (3.9) | 12.5 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Amenorrhea
Description: Amenorrhea was defined as menstrual blood loss (MBL) < 2 mL during the last 28 days of treatment. The evaluation of MBL was based on the Alkaline hematin (AH) method.
Time Frame: The last 28 days of treatment period 1
Population: FAS population with evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 32 | 33 | 31
Participants | 29 | 1 | 25
Statistical Analysis 1: Comparison: Vilaprisan (A1) vs Placebo+Vilaprisan (B1) vs Vilaprisan+Placebo (B2); Vilaprisan (A1) and Vilaprisan+Placebo (B2) combined vs. Placebo+Vilaprisan (B1) in treatment period 1; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.82, 95% CI 2-sided [0.72 to 0.93] — Number of subjects per treatment: 63 (Vilaprisan) / 33 (Placebo)

2. Secondary Outcome: Number of Participants With Heavy Menstrual Bleeding (HMB) Response
Description: HMB was defined as MBL <80.00 mL during the last 28 days of treatment and >50% reduction compared to baseline (assessed by the AH method).
Time Frame: The last 28 days of treatment period 1 and treatment period 2
Population: FAS population with valuable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 32 | 33 | 31
Participants
  Treatment period 1 | 30 | 7 | 26
  Treatment period 2: number analyzed (Participants) | 8 | 10 | 8
  Treatment period 2 | 6 | 9 | 1

3. Secondary Outcome: Time to Onset of Amenorrhea
Description: Onset of amenorrhea was defined by the first day for which the MBL for all subsequent 28-day periods up to the end of a treatment period was <2 mL (amenorrhea defined similar to primary endpoint and assessed by the AH method).
Time Frame: In treatment period 1 (12 weeks) and in treatment period 2 (12 weeks)
Population: FAS population with valuable data. In treatment period 2, participants who did not start the respective treatment period or had less than 28 days of treatment are included among censored observations.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 32 | 33 | 31
Days
  Treatment period 1 | 3 [2 to 4] | NA [NA to NA] — NA: value could not be estimated due to censored data. | 3 [1 to 9]
  Treatment period 2: number analyzed (Participants) | 8 | 10 | 8
  Treatment period 2 | 3 [2 to 20] | 4 [3 to NA] — NA: value could not be estimated due to censored data. | NA [NA to NA] — NA: value could not be estimated due to censored data.

4. Secondary Outcome: Time to Onset of Controlled Bleeding
Description: Onset of controlled bleeding was defined by the first day for which the MBL for all subsequent 28-day periods up to the end of a treatment period was <80.00 mL (assessed by the AH method).
Time Frame: In treatment period 1 (12 weeks) and in treatment period 2 (12 weeks)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 32 | 33 | 31
Days
  Treatment period 1 | 1 [1 to 1] | NA [NA to NA] — NA: value could not be calculated because less than 50% of subjects in group showed response. | 1 [1 to 2]
  Treatment period 2: number analyzed (Participants) | 8 | 10 | 8
  Treatment period 2 | 1.5 [1 to 1.9] | 1 [1 to 2] | NA [NA to NA] — NA: value could not be calculated because less than 50% of subjects in group showed response.

5. Secondary Outcome: Number of Participants With Absence of Bleeding (Spotting Allowed)
Description: Absence of bleeding was defined as no scheduled or unscheduled bleeding (spotting allowed) during the last 28 days of a treatment period based on subjects' daily responses to the UF-DBD (Uterine Fibroid Daily Bleeding Diary).
Time Frame: The last 28 days of treatment period 1 and treatment period 2
Population: FAS population with valuable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 32 | 33 | 31
Participants
  Treatment period 1 | 29 | 2 | 25
  Treatment period 2: number analyzed (Participants) | 8 | 10 | 8
  Treatment period 2 | 6 | 8 | 1

6. Secondary Outcome: Number of Participants by Endometrial Biopsy Main Results (Majority Read, Main Diagnosis)
Description: Number of participants with endometrial histology findings, e.g. benign endometrium, malignant neoplasm, hyperplasia without atypia, hyperplasia with atypia and endometrial polyps.
Time Frame: Up to 36 weeks
Population: Samples with sufficient tissue for analysis in SAF population was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 31 | 30 | 30
Participants
  Adequate endometrial tissue: number analyzed (Participants) | 31 | 30 | 29
  Adequate endometrial tissue | 31 | 30 | 26
  Benign Endometrium: number analyzed (Participants) | 31 | 30 | 29
  Benign Endometrium | 31 | 30 | 26
  Hyperplasia WHO 2014, no atypia: number analyzed (Participants) | 31 | 30 | 29
  Hyperplasia WHO 2014, no atypia | 0 | 0 | 0
  Hyperplasia WHO 2014, atypia: number analyzed (Participants) | 31 | 30 | 29
  Hyperplasia WHO 2014, atypia | 0 | 0 | 0
  Malignant Neoplasm: number analyzed (Participants) | 31 | 30 | 29
  Malignant Neoplasm | 0 | 0 | 0
  Endometrial Polyps: number analyzed (Participants) | 31 | 30 | 29
  Endometrial Polyps | 2 | 0 | 1

7. Secondary Outcome: Change From Baseline of Endometrial Thickness
Description: Ultrasound examinations were performed. Endometrial thickness was measured in the medio-sagittal section as double-layer in millimeters. Summary statistics for change from baseline in endometrial thickness was provided in below table.
Time Frame: In treatment period 1 (12 weeks) and in treatment period 2 (12 weeks)
Population: SAF was analyzed. Overall number of participants analyzed represents number of participants without missing data.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Vilaprisan (A1) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 31 | 30 | 30
Millimeters
  Treatment period 1: number analyzed (Participants) | 30 | 30 | 29
  Treatment period 1 | -2.5 (4.1) | -2.8 (2.6) | -3.1 (3.7)
  Treatment period 2: number analyzed (Participants) | 7 | 10 | 7
  Treatment period 2 | -5.3 (7.6) | -3.5 (4.1) | -0.4 (4.1)

ADVERSE EVENTS:
Time Frame: For TEAEs: started from the first application of study medication up to 60 calendar days after end of treatment with study medication. For Post-treatment AEs: started from Day 61 after the end of treatment with study medication (All AEs identified during the safety follow-up are included in this portion).
Groups:
- Vilaprisan (A1) - Treatment Emergent AEs: Vilaprisan in treatment period 1 for 12 weeks and in treatment period 2 for 12 weeks, separated by 1 bleeding episode. TEAEs: defined as AEs that "started from the first application of study medication up to 60 calendar days after end of treatment with study medication".
- Placebo+Vilaprisan (B1) - Treatment Emergent AEs: Placebo in treatment period 1 for 12 weeks, and vilaprisan in treatment period 2 for 12 weeks, separated by 1 bleeding episode. TEAEs: defined as AEs that "started from the first application of study medication up to 60 calendar days after end of treatment with study medication".
- Vilaprisan +Placebo (B2) - Treatment Emergent AEs: Vilaprisan in treatment period 1 for 12 weeks, and placebo in treatment period 2 for 12 weeks, separated by 1 bleeding episode. TEAEs: defined as AEs that "started from the first application of study medication up to 60 calendar days after end of treatment with study medication".
- Vilaprisan (A1) - Post Treatment AEs: Vilaprisan in treatment period 1 for 12 weeks and in treatment period 2 for 12 weeks, separated by 1 bleeding episode. Post-treatment AEs: defined as all AEs that started from Day 61 after the end of treatment with study medication. (All AEs identified during the safety follow-up are included in this portion).
- Placebo+Vilaprisan (B1) - Post Treatment AEs: Placebo in treatment period 1 for 12 weeks, and vilaprisan in treatment period 2 for 12 weeks, separated by 1 bleeding episode. Post-treatment AEs: defined as all AEs that started from Day 61 after the end of treatment with study medication. (All AEs identified during the safety follow-up are included in this portion).
- Vilaprisan+Placebo (B2) - Post Treatment AEs: Vilaprisan in treatment period 1 for 12 weeks, and placebo in treatment period 2 for 12 weeks, separated by 1 bleeding episode. Post-treatment AEs: defined as all AEs that started from Day 61 after the end of treatment with study medication. (All AEs identified during the safety follow-up are included in this portion).
Arm/Group | Vilaprisan (A1) - Treatment Emergent AEs | Placebo+Vilaprisan (B1) - Treatment Emergent AEs | Vilaprisan +Placebo (B2) - Treatment Emergent AEs | Vilaprisan (A1) - Post Treatment AEs | Placebo+Vilaprisan (B1) - Post Treatment AEs | Vilaprisan+Placebo (B2) - Post Treatment AEs
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/30 | 0/31 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/31 | 4/30 | 0/30 | 7/31 | 8/30 | 3/30
Other Adverse Events (participants affected / at risk) | 18/31 | 19/30 | 16/30 | 10/31 | 12/30 | 12/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilaprisan (A1) - Treatment Emergent AEs (N=31) | Placebo+Vilaprisan (B1) - Treatment Emergent AEs (N=30) | Vilaprisan +Placebo (B2) - Treatment Emergent AEs (N=30) | Vilaprisan (A1) - Post Treatment AEs (N=31) | Placebo+Vilaprisan (B1) - Post Treatment AEs (N=30) | Vilaprisan+Placebo (B2) - Post Treatment AEs (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Myomectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Salpingectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary cystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hysterosalpingectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uterine dilation and curettage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometriosis ablation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma embolisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilaprisan (A1) - Treatment Emergent AEs (N=31) | Placebo+Vilaprisan (B1) - Treatment Emergent AEs (N=30) | Vilaprisan +Placebo (B2) - Treatment Emergent AEs (N=30) | Vilaprisan (A1) - Post Treatment AEs (N=31) | Placebo+Vilaprisan (B1) - Post Treatment AEs (N=30) | Vilaprisan+Placebo (B2) - Post Treatment AEs (N=30)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 4 (4) | 5 (9) | 1 (1) | 5 (5)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (3)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (2) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Premenstrual syndrome (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial thickening (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hot flush (Vascular disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
* The trial was terminated earlier than planned. It was sufficiently advanced to allow for meaningful analysis.
* In many subjects, follow up phase was longer than the planned one.
* Safety evaluations were not limited to the planned timepoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT03400956/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT03400956/SAP_001.pdf